CLINICAL TRIAL: NCT05885646
Title: Treatment of Epilepsy Syndromes of Childhood With Sleep Activation Using Sulthiame: an Exploratory Study of the Short Term Effect on EEG
Brief Title: Effect of Sulthiame on EEG in Childhood Epilepsy Syndromes
Acronym: SURF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC23_0073
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Importance of Interictal Epileptiform Activity on Sleep EEG; Epilepsy in Children
MeSH Terms: interventions — sulthiame

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Sulthiame — Sulthiame add-on according to good clinical practice in these childhood epilepsy syndromes

SUMMARY:
The effect of sulthiame on EEG has been studied in epilepsy syndromes of childhood with sleep activation by comparing sleep EEG obtained at baseline and after 4 weeks of treatment. The aim of the study is to know if an effect is still identifiable after 2 weeks of treatment by performing sleep EEG recordings after 2 and 4 weeks of treatment, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy syndromes of childhood with sleep activation
* Failure of at least two anti-epileptic drugs (AED)
* Sleep EEG performed in the last 7 days before inclusion and showing interictal epileptiform discharges (baseline EEG)

Exclusion Criteria:

* Previous trial with sulthiame
* More than 2 AED at inclusion
* Use of corticosteroids at inclusion
* Change in the anti-epileptic treatment in the 7 days before baseline EEG

Ages: 6 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: -Children with pharmaco-resistant epilepsy
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients showing improved sleep EEG at day 14 compared to baseline EEG | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Van Bogaert, Professor, Principal Investigator — Angers University Hospital
Locations (3):
- France (3):
  - Angers University Hospital, Pediatric department, Angers
  - Strasbourg University Hospital, Pediatric department, Strasbourg
  - Toulouse University Hospital, Pediatric Neurology Department, Toulouse

IPD SHARING:
Plan to Share IPD: No